CLINICAL TRIAL: NCT05833139
Title: The Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of a Single Oral Dose of BI 1810631 in Healthy Male Subjects (an Open-label, Two-period, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of Zongertinib (BI 1810631) in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0004; 2022-003757-63 (EudraCT Number)
Record Dates: First submitted 2023-02-28; First posted 2023-04-27 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zongertinib alone (R) / Zongertinib + itraconazole (T) (Experimental): Treatment Period 1: a single oral dose of 15 milligrams (mg) zongertinib, film-coated tablet, was administered once on Day 1 (Day 1, Period 1, Visit 2), as reference treatment R.
  Treatment Period 2: a single oral solution of 200 mg (10 mg/mL in a 20 milliliter (mL) solution) itraconazole was administered once daily over 14 days ([total: 14 doses], from Day -3 to Day 11, Period 2). On Day 1 (Day 1, Period 2, Visit 3), 4th day of itraconazole treatment, a single oral dose of 15 mg zongertinib was administered 1 hour (h) after itraconazole administration as test treatment T.
  The two administrations of zongertinib were separated by a washout interval of at least 14 days.
  Zongertinib and itraconazole were orally administered with 240 mL of water after an overnight fast of at least 10 h for zongertinib and 9 h for itraconazole.
  Interventions: Drug: Zongertinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Zongertinib — Zongertinib
  Other Names: BI 1810631, Hernexeos®
Drug: Itraconazole — Itraconazole
  Other Names: Sempera® Liquid

SUMMARY:
The main objective of this trial is to investigate the effect of multiple doses of the strong CYP3A inhibitor and recommended P-glycoprotein (P-gp) inhibitor itraconazole on the pharmacokinetics of a single dose of zongertinib in plasma following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomised, open-label, two-treatment, two-period, fixed-sequence crossover trial in healthy men. There was one group of participants, each participant underwent the fixed sequence of Reference (R) followed by Test (T) treatment, with a washout period of ≥14 days between zongertinib (BI 1810631) administrations.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Study Period 1
Arm/Group | Zongertinib Alone (R) / Zongertinib + Itraconazole (T)
Started | 16
Completed | 16
Not Completed | 0
Period: Study Period 2
Arm/Group | Zongertinib Alone (R) / Zongertinib + Itraconazole (T)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all participants who were treated with at least one dose of trial drug. The treated set was used for the safety analyses.
Arm/Group | Zongertinib Alone (R) / Zongertinib + Itraconazole (T)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of zongertinib in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: Within 3 hours (h) prior to, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34, 47, 71, 119, 167 h for both periods, and additionally at 191, 215, 239, 263, and 287 h for period 2, after zongertinib administration.
Population: Pharmacokinetic (PK) Set (PKS): this set included all participants in the treated set (TS) who provided at least one primary or secondary PK endpoint, and who was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles * hour per Liter
Groups:
- Zongertinib Alone: Treatment Period 1: a single oral dose of 15 milligrams (mg) zongertinib, film-coated tablet, was administered once on Day 1 (Day 1, Period 1, Visit 2) with 240 mL of water after an overnight fast of at least 10 hours (h).
- Zongertinib + Itraconazole: Treatment Period 2: a single oral solution of 200 mg itraconazole (10 mg/mL in a 20 mL solution) was administered once daily over 14 days ([total: 14 doses], from Day -3 to Day 11, Period 2). On Day 1, of the itraconazole treatment (Day 1, Period 2, Visit 3), a single oral dose of 15 mg zongertinib was administered 1 h after itraconazole administration.
Arm/Group | Zongertinib Alone | Zongertinib + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles * hour per Liter | 3014 (NA) — Adjusted Geometric Standard Error = 1.068 | 4255 (NA) — Adjusted Geometric Standard Error = 1.068
Statistical Analysis 1: Comparison: Zongertinib Alone vs Zongertinib + Itraconazole; The statistical model used was an analysis of variance (ANOVA) on the logarithmic scale. AUC0-∞ was log transformed (natural logarithm) prior to fitting the ANOVA model, considering the effect 'participant' as random and "treatment" as fixed; Test type: Other; ANOVA; Geometric mean ratio (T/R) [%] = 141.2, 90% CI 2-sided [126.3 to 157.7] — Intra-individual geometric coefficient of variation (gCV%) = 18.0

2. Primary Outcome: Maximum Measured Concentration of Zongertinib in Plasma (Cmax)
Description: Maximum measured concentration of zongertinib in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: PKS: this set included all participants in the TS who provided at least one primary or secondary PK endpoint, and who was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles per Liter
Arm/Group | Zongertinib Alone | Zongertinib + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles per Liter | 138 (NA) — Adjusted Geometric Standard Error = 1.094 | 175 (NA) — Adjusted Geometric Standard Error = 1.094
Statistical Analysis 1: Comparison: Zongertinib Alone vs Zongertinib + Itraconazole; The statistical model used was an analysis of variance (ANOVA) on the logarithmic scale. Cmax was log transformed (natural logarithm) prior to fitting the ANOVA model, considering the effect 'participant' as random and "treatment" as fixed; Test type: Other; ANOVA; Geometric mean ratio (T/R) [%] = 126.9, 90% CI 2-sided [106.6 to 151.0] — Intra-individual geometric coefficient of variation (gCV%) = 28.7

3. Secondary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of zongertinib in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles * hour per Liter
Arm/Group | Zongertinib Alone | Zongertinib + Itraconazole
Number analyzed (Participants) | 16 | 16
Nanomoles * hour per Liter | 2892 (NA) — Adjusted Geometric Standard Error = 1.071 | 4130 (NA) — Adjusted Geometric Standard Error = 1.071
Statistical Analysis 1: Comparison: Zongertinib Alone vs Zongertinib + Itraconazole; The statistical model used was an analysis of variance (ANOVA) on the logarithmic scale. AUC0-tz was log transformed (natural logarithm) prior to fitting the ANOVA model, considering the effect 'participant' as random and "treatment" as fixed; Test type: Other; ANOVA; Geometric mean ratio (T/R) [%] = 142.8, 90% CI 2-sided [126.0 to 161.9] — Intra-individual geometric coefficient of variation (gCV%) = 20.4

ADVERSE EVENTS:
Time Frame: Zongertinib alone: From the first administration of zongertinib until first administration of itraconazole (IT), up to 14 days. IT alone: From the first administration of itraconazole until 2nd administration of zongertinib, up to 3 days. Zongertinib + IT: From the second administration of zongertinib until 8 days after the last administration of IT, up to 19 days.
Description: Treated Set (TS): this set included all participants who were treated with at least one dose of trial drug. The TS was used for safety analyses.
Groups:
- Itraconazole Alone: Treatment period 2: a single oral dose of 200 mg itraconazole (10 mg/milliliter (mL) in a 20 mL solution) was administered once daily with 240 mL of water after an overnight fast of 9 hours (h) over 3 days ([total: 3 doses], from Day -3 to Day -1, Period 2, Visit 3).
- Zongertinib + Itraconazole: Treatment Period 2: a single oral solution of 200 mg itraconazole (10 mg/mL in a 20 mL solution) was administered once daily over 11 days ([total: 11 doses], from Day 1 to Day 11, Period 2). On Day 1, of the itraconazole treatment (Day 1, Period 2, Visit 3), a single oral dose of 15 mg zongertinib was administered 1h after itraconazole administration.
Arm/Group | Zongertinib Alone | Itraconazole Alone | Zongertinib + Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 6/16 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zongertinib Alone (N=16) | Itraconazole Alone (N=16) | Zongertinib + Itraconazole (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT05833139/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05833139/SAP_001.pdf